CLINICAL TRIAL: NCT01131858
Title: A Placebo Controlled Double Blinded Study of Vitamin D3 Substitution to Patients With Primary Immunodeficiency
Brief Title: Study of Vitamin D3 Substitution to Patients With Primary Immunodeficiency
Acronym: VITAPID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Peter Bergman, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009/1678-31/4
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Primary Immune Deficiency Disorder
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Vitamin D (Active Comparator): Vigantol (cholecalciferol) 4000 IE/day
  Interventions: Drug: Vigantol

INTERVENTIONS:
Drug: Vigantol — Vigantol 4000IU/day
  Arms: Vitamin D
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Hypothesis: Cholecalciferol (vitamin D3) prevent respiratory tract infections in patients with primary immunodeficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Increased number of respiratory tract infections
* At least 42 days of infections during 2008 or 2009
* S-25 OH vitamin D3 < 250 nM
* Not planning a pregnancy during the coming year
* Accepting the use of contraceptives during 1 year

Exclusion Criteria:

* Continuous antibiotic treatment
* Hypercalcemia
* Sarcoidosis
* Kidney disease
* Tuberculosis
* Pregnancy
* Kidney stone
* Heart medication (glycosides)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Infectious score | 12 months

SECONDARY OUTCOMES:
Antimicrobial peptide expression in nasal fluid | 12 months
Serum levels of 25-OH Vitamin D3 | 12 months
Consumption of antibiotics | 12 months
Number of positive bacterial cultures in nasal swabs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Andersson, MD/PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska Univerisity Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Bergman P, Norlin AC, Hansen S, Bjorkhem-Bergman L. Vitamin D supplementation improves well-being in patients with frequent respiratory tract infections: a post hoc analysis of a randomized, placebo-controlled trial. BMC Res Notes. 2015 Sep 29;8:498. doi: 10.1186/s13104-015-1504-2. PMID 26419363
- [Derived] Bergman P, Norlin AC, Hansen S, Bjorkhem-Bergman L. Vitamin D supplementation to patients with frequent respiratory tract infections: a post hoc analysis of a randomized and placebo-controlled trial. BMC Res Notes. 2015 Aug 30;8:391. doi: 10.1186/s13104-015-1378-3. PMID 26319134